CLINICAL TRIAL: NCT02964286
Title: The Effect of Acupoint Massotherapy on Relieving Chemotherapy-induced Myelosupression Among Patients With Cancer
Brief Title: The Effect of Acupoint Massotherapy on Relieving Chemotherapy-induced Myelosupression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TMU-JIRB: 201501030
Record Dates: First submitted 2016-10-31; First posted 2016-11-16 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-07

CONDITIONS: Cancer, Breast; Acupressure; Hematopoiesis
Keywords: Cancer; Acupressure; Hematopoietic Cell Growth Factors
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupressure group (Experimental): The intervention technique used is ''The electric vibrating massager'', ''SAMPO®'', and patients are taught to apply the strong mode on the 15 specific points,5 min each, 3 times a day from Monday to Friday during chemotherapy course. The intervention follows the points are used to stimulate the hematopoietic function. including Hegu (LI4), Quchi (LI11), Xuehai (SP10); Sanyin-jiao (SP6), Taixi (K3), Zusanli (ST36), Taichong (LV3), Baihui (GV20). Before the study, the trained study nurses teach patients that how to use the technique and stuck adhesive dots label on each specific acupoints.
  Interventions: Device: The Electric vibrating massager,SAMPO®
- Control group (No Intervention): The patients of the control group are not admitted any acupoints press-related interventions, only take clinical treatment protocol as usual.

INTERVENTIONS:
Device: The Electric vibrating massager,SAMPO® — The technique used is The electric vibrating massager ''SAMPO®'', and patients are taught to apply the strong mode on the 15 specific points,5 min each, 3 times a day from Monday to Friday during chemotherapy course. The intervention follow the points are used to stimulate the hematopoietic function. According to their anatomical location: upper extremity are Hegu (LI4), Quchi (LI11); lower extremity are Xuehai (SP10); Sanyin-jiao (SP6), Taixi (K3), Zusanli (ST36), Taichong (LV3); and the top of head is Baihui (GV20). The used of all the points, except for Baihui (GV20), is bilateral.
  Arms: Acupressure group

SUMMARY:
In this proposed project, the investigator will estimate the effect of massotherapy of acupoints on alleviating chemotherapy-induced myelosuppression among patients with cancer.

DETAILED DESCRIPTION:
Chemotherapy is mainly used to treat and control the progression of gynecological cancer, bone marrow suppression the evil side effects after chemotherapy, which may decreasing immune function and further causes serious fatal infections.

Acupuncture is a valid intervention in medical practice and has been used for the improvement of chemotherapy-induced leucopenia. In a systematic meta-analysis study showed that acupoints stimulation has immunomodulatory effect for therapy induced bone marrow suppression in cancer patients. Therefore, in the acupressure group, the technique used is the electric vibrating massager, and patients are taught to apply the strong mode on the 15 specific points,5 min each, 3 times a day during chemotherapy.The intervention follows the points are used to stimulate the hematopoietic function including Hegu (LI4), Quchi (LI11), Xuehai (SP10); Sanyin-jiao (SP6), Taixi (K3), Zusanli(ST36), Taichong (LV3); and Baihui (GV20). The patients of the control group are not admitted any acupoints press-related interventions mentioned above.

The purpose of this study is to evaluate the effectiveness of non-invasive acupressure on the prevention of chemotherapy-induced myelosuppression among patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed of gynecologic cancer, regardless of stage.
* receiving initial chemotherapy.
* ability to write informed consent.
* between 20 to 70 years old.

Exclusion Criteria:

* history of severe cardiac disorder.
* suffering from the hematological diseases such as hemolytic anemia.
* cancer patients with lymphoedema at the area of the acupressure points.
* diagnosed combine with other cancers.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The Effect of Acupoint Massotherapy on Relieving Chemotherapy-induced Myelosuppression Among Patients With Cancer. | Two years
  To evaluate the effectiveness and mechanisms of acupressure in the prevention and diminishing of chemotherapy-induced myelosuppression among patients with gynecologic cancer.
  Using a composite outcome measure consisting of blood counts and plasma. Blood counts: white blood cells, platelets, hemoglobin and red blood cells.
  Plasma: Stem cell factor(SCF)、Granulocyte-macrophage colony-stimulating factor(GM-CSF)、Interleukin-1(IL-1)、 Interleukin-2(IL-2)、Interleukin-3 (IL-3)、Interleukin-6(IL-6)、Interleukin-8(IL-8)、Interleukin-12(IL-12)、Transforming growth factor-B (TGF-B)、Interferon gamma(IFN-r)、Tumor necrosis factor-a(TNF-a)

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu-Ting Tsai, PhD, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wen CP, Wai JP, Tsai MK, Yang YC, Cheng TY, Lee MC, Chan HT, Tsao CK, Tsai SP, Wu X. Minimum amount of physical activity for reduced mortality and extended life expectancy: a prospective cohort study. Lancet. 2011 Oct 1;378(9798):1244-53. doi: 10.1016/S0140-6736(11)60749-6. Epub 2011 Aug 16. PMID 21846575
- [Result] Goh J, Kirk EA, Lee SX, Ladiges WC. Exercise, physical activity and breast cancer: the role of tumor-associated macrophages. Exerc Immunol Rev. 2012;18:158-76. PMID 22876727
- [Result] Mason C, Alfano CM, Smith AW, Wang CY, Neuhouser ML, Duggan C, Bernstein L, Baumgartner KB, Baumgartner RN, Ballard-Barbash R, McTiernan A. Long-term physical activity trends in breast cancer survivors. Cancer Epidemiol Biomarkers Prev. 2013 Jun;22(6):1153-61. doi: 10.1158/1055-9965.EPI-13-0141. Epub 2013 Apr 10. PMID 23576689
- [Result] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Result] Singh AA, Jones LW, Antonelli JA, Gerber L, Calloway EE, Shuler KH, Freedland SJ, Grant DJ, Hoyo C, Banez LL. Association between exercise and primary incidence of prostate cancer: does race matter? Cancer. 2013 Apr 1;119(7):1338-43. doi: 10.1002/cncr.27791. Epub 2013 Feb 11. PMID 23401030
- [Result] Behrens G, Matthews CE, Moore SC, Freedman ND, McGlynn KA, Everhart JE, Hollenbeck AR, Leitzmann MF. The association between frequency of vigorous physical activity and hepatobiliary cancers in the NIH-AARP Diet and Health Study. Eur J Epidemiol. 2013 Jan;28(1):55-66. doi: 10.1007/s10654-013-9767-1. Epub 2013 Jan 26. PMID 23354983
- [Result] Santoso JT, Crigger M, English E, Wan J, Likes W. Smoking cessation counseling in women with genital intraepithelial neoplasia. Gynecol Oncol. 2012 Jun;125(3):716-9. doi: 10.1016/j.ygyno.2012.02.018. Epub 2012 Feb 21. PMID 22366589
- [Result] Lee IM, Shiroma EJ, Lobelo F, Puska P, Blair SN, Katzmarzyk PT; Lancet Physical Activity Series Working Group. Effect of physical inactivity on major non-communicable diseases worldwide: an analysis of burden of disease and life expectancy. Lancet. 2012 Jul 21;380(9838):219-29. doi: 10.1016/S0140-6736(12)61031-9. PMID 22818936
- [Result] Wu Y, Zhang D, Kang S. Physical activity and risk of breast cancer: a meta-analysis of prospective studies. Breast Cancer Res Treat. 2013 Feb;137(3):869-82. doi: 10.1007/s10549-012-2396-7. Epub 2012 Dec 30. PMID 23274845
- [Result] Lu W, Matulonis UA, Doherty-Gilman A, Lee H, Dean-Clower E, Rosulek A, Gibson C, Goodman A, Davis RB, Buring JE, Wayne PM, Rosenthal DS, Penson RT. Acupuncture for chemotherapy-induced neutropenia in patients with gynecologic malignancies: a pilot randomized, sham-controlled clinical trial. J Altern Complement Med. 2009 Jul;15(7):745-53. doi: 10.1089/acm.2008.0589. PMID 19552597
- [Result] Ye F, Chen S, Liu W. Effects of electro-acupuncture on immune function after chemotherapy in 28 cases. J Tradit Chin Med. 2002 Mar;22(1):21-3. PMID 11977512
- [Result] Ye F, Liu D, Wang S, Xu L. Effects of electro-acupuncture on T cell subpopulations, NK activity, humoral immunity and leukocyte count in patients undergoing chemotherapy. J Tradit Chin Med. 2007 Mar;27(1):19-21. PMID 17393618
- [Result] Han YF, Gong Z, Huang LQ, Xia X, Zhao WJ. [Clinical study on acupuncture for leukopenia induced by chemotherapy]. Zhongguo Zhen Jiu. 2010 Oct;30(10):802-5. Chinese. PMID 21058473
- [Result] Raghavendran HR, Sathyanath R, Shin J, Kim HK, Han JM, Cho J, Son CG. Panax ginseng modulates cytokines in bone marrow toxicity and myelopoiesis: ginsenoside Rg1 partially supports myelopoiesis. PLoS One. 2012;7(4):e33733. doi: 10.1371/journal.pone.0033733. Epub 2012 Apr 16. PMID 22523542
- [Result] Jong MS, Hwang SJ, Chen FP. Effects of electro-acupuncture on serum cytokine level and peripheral blood lymphocyte subpopulation at immune-related and non-immune-related points. Acupunct Electrother Res. 2006;31(1-2):45-59. doi: 10.3727/036012906815844337. PMID 17063830
- [Result] Joos S, Schott C, Zou H, Daniel V, Martin E. Immunomodulatory effects of acupuncture in the treatment of allergic asthma: a randomized controlled study. J Altern Complement Med. 2000 Dec;6(6):519-25. doi: 10.1089/acm.2000.6.519. PMID 11152056
- [Result] Gautam A, Bepler G. Suppression of lung tumor formation by the regulatory subunit of ribonucleotide reductase. Cancer Res. 2006 Jul 1;66(13):6497-502. doi: 10.1158/0008-5472.CAN-05-4462. PMID 16818620
- [Result] Tsai HT, Su PH, Lee TH, Tee YT, Lin LY, Yang SF, Wang PH. Significant elevation and correlation of plasma neutrophil gelatinase associated lipocalin and its complex with matrix metalloproteinase-9 in patients with pelvic inflammatory disease. Clin Chim Acta. 2011 Jun 11;412(13-14):1252-6. doi: 10.1016/j.cca.2011.03.021. Epub 2011 Mar 23. PMID 21439274